CLINICAL TRIAL: NCT02426996
Title: Treatment of Chronic Anterior Shoulder Instability by a Latarjet-type Bone Block Procedure Using the SEM (Science Et Medecine) Positioning Tool: Using a Scan to Assess Consolidation and Return to Normal Activity at 3 Months
Brief Title: The Latarjet-type Procedure Using the SEM Positioner: Using a Scan to Assess Consolidation
Acronym: IACE Scan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting patients difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2014/OM-01; 2015-A00155-44 (Other: RCB number)
Record Dates: First submitted 2015-04-15; First posted 2015-04-27 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2017-08

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study population (Experimental): The patients included have been operated for chronic anterior shoulder instability by a Latarjet-type bone block procedure using the SEM (Science Et Medecine) positioning tool within the past 3 months.
  Intervention: Scan of shoulder
  Interventions: Procedure: Scan of shoulder

INTERVENTIONS:
Procedure: Scan of shoulder — A scan (no injection) of the concerned shoulder will be performed at 3 months post-surgery. Cuts in three planes of space, including all of the glenoid. 3D reconstructions.

SUMMARY:
The main objective of this study is to evaluate, after surgery for chronic anterior shoulder instability using a Latarjet technique with positioning of the bone block via an SEM positioning tool, the value of the contribution of a shoulder scan at 3 months post surgery in the decision to return to activity early as conditioned by the quality of the bone block consolidation.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess:

A. the position of the block according to a shoulder scan at 3 months post-surgery

B. functional scores (Constant, Walch-Duplay) at 6 weeks, 3 and 6 months post surgery.

C. Complications: osteoarthritis, lysis of the block.

D. pain.

E. date of return to full activity.

F. patient satisfaction concerning care (visual analog scale at 6 months post-surgery).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient was operated for chronic anterior shoulder instability (defined by a history of at least two true dislocations and an ISIS score> 2) 6 weeks ago (+/- 5 days)

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Did the patient return to activity at 3 months? yes/no | Week 6 after inclusion, which = 3 months after surgery

SECONDARY OUTCOMES:
Constant score | week -6
Constant score | day 0 (study inclusion)
Constant score | week 6
Constant score | week 18
Walch-Duplay score | week -6
Walch-Duplay score | day 0 (study inclusion)
Walch-Duplay score | week 6
Walch-Duplay score | week 18
Presence/absence of complications | day 0 (study inclusion)
Presence/absence of complications | week 6
Presence/absence of complications | week 18
Visual analog scale for pain | day 0 (study inclusion)
Visual analog scale for pain | week 6
Visual analog scale for pain | week 18
Date of return to total activity | week 18
Visual analog scale for satisfaction | week 18

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marès, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Clinique Saint Jean, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes